CLINICAL TRIAL: NCT00005118
Title: A Multicenter, Open-Label, 24-Week Study to Evaluate the Efficacy and Safety of Indinavir Sulfate 800 Mg and Ritonavir 200 Mg b.i.d. Plus 2 NRTIs b.i.d. in HIV-1 Infected Individuals Who Require Early Treatment Intervention
Brief Title: The Safety and Effectiveness of Indinavir Plus Ritonavir Plus Two NRTIs in HIV-Infected Patients Who Need Early Intervention Treatment
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Merck Sharp & Dohme LLC (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 246V; CRX481; 107-00
Record Dates: First submitted 2000-04-07; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2001-07

CONDITIONS: HIV Infections
Keywords: HIV-1; Drug Therapy, Combination; HIV Protease Inhibitors; Ritonavir; Indinavir; Reverse Transcriptase Inhibitors; Anti-HIV Agents; Viral Load; Nelfinavir
MeSH Terms: conditions — HIV Infections | interventions — Indinavir; Ritonavir

INTERVENTIONS:
Drug: Indinavir sulfate
Drug: Ritonavir

SUMMARY:
The purpose of this study is to see if it is safe and effective to give indinavir plus ritonavir plus 2 NRTIs to HIV-infected patients who need early intervention treatment.

DETAILED DESCRIPTION:
Patients receive indinavir bid plus ritonavir bid, plus 2 NRTIs bid (2 new NRTIs or 1 new NRTI and 1 NRTI without evidence of resistance). CD4 cell counts and plasma viral RNA are measured every 4 weeks for the duration of the study. Physical examination and laboratory tests of blood and urine are performed every 4 weeks for the duration of the study. Chest x-ray and 12-lead ECG are done prestudy.

ELIGIBILITY:
Inclusion Criteria

Patients may be eligible for this study if they:

* Are HIV-positive.
* Are 18 years of age or older.
* Have a CD4 cell count of at least 50 cells/mm3.
* Have a viral load (level of HIV in the blood) of at least 400 copies/ml but no more than 20,000 copies/ml.
* Have had an initial response to protease inhibitor therapy with a viral load of less than 400 copies/ml in two consecutive tests at least 1 week apart.
* Have been on anti-HIV (antiretroviral) treatment including indinavir or nelfinavir for at least 16 weeks.
* Have had virologic failure (two consecutive viral loads that were greater than or equal to 400 copies/ml and less than or equal to 20,000 copies/ml at least 1 week apart) that is not due to another infection, vaccination, or a temporary stop in treatment.
* Are naive to at least one of the selected NRTIs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100

CONTACTS AND LOCATIONS:
Locations (40):
- United States (40):
  - Pacific Oaks Research, Beverly Hills, California
  - Ocean View Internal Medicine, Long Beach, California
  - Bisher Akil, Los Angeles, California
  - Tower Infectious Diseases / Med Associates Inc, Los Angeles, California
  - UCSD Med Ctr - Owen Clinic, San Diego, California
  - HIV Institute / Davies Med Ctr, San Francisco, California
  - San Francisco Veterans Adm Med Cntr, San Francisco, California
  - Avalar Medical Group, Tarzana, California
  - Harbor - UCLA Med Ctr, Torrance, California
  - Benjamin Young, Denver, Colorado
  - University of Connecticut Health Center, Farmington, Connecticut
  - IDC Research Initiative, Altamonte Springs, Florida
  - Hillsborough County Health Dept, Tampa, Florida
  - Mercer University School of Medicine, Macon, Georgia
  - Thomas Coffman MD, Boise, Idaho
  - Chicago Ctr for Clinical Research, Chicago, Illinois
  - Northwestern Univ / Infect Dis Div / Pasavant Pav 828, Chicago, Illinois
  - The CORE Ctr, Chicago, Illinois
  - Univ of Kansas School of Medicine, Wichita, Kansas
  - University of Louisville / ID Division, Louisville, Kentucky
  - Tulane Univ School of Medicine, New Orleans, Louisiana
  - Institute of Human Virology, Baltimore, Maryland
  - New England Med Ctr, Boston, Massachusetts
  - Cooper Hospital Early Intervention Program, Camden, New Jersey
  - Dr Ronald Nahass, Somerville, New Jersey
  - Mt Vernon Hosp, Mount Vernon, New York
  - Gramercy Park Physicians LLP, New York, New York
  - St Luke Roosevelt Hosp, New York, New York
  - St Vincents Hosp / Clinical Research Program, New York, New York
  - Bellevue Hosp Ctr, New York, New York
  - Mount Sinai Med Ctr, New York, New York
  - SUNY at Stony Brook / Div of Infectious Disease, Stony Brook, New York
  - Bronx Veterans Affairs Med Ctr, The Bronx, New York
  - Wake Forest Univ School of Medicine, Winston-Salem, North Carolina
  - Oklahoma Univ Health Science Ctr, Oklahoma City, Oklahoma
  - Fanno Creek Clinic, Portland, Oregon
  - Anderson Clinical Research, Pittsburgh, Pennsylvania
  - Univ of Texas Med Branch / Div of Infectious Dis, Galveston, Texas
  - Thomas Street Clinic, Houston, Texas
  - Univ of Texas Health Sciences Ctr, San Antonio, Texas